CLINICAL TRIAL: NCT05527158
Title: The Impact of Traditional Chinese Yijinjing Exercise on Hand Dysfunction in Rheumatoid Arthritis Patients:a Randomized Controlled Trial Protocol
Brief Title: Traditional Chinese Yijinjing Exercise on Hand Dysfunction in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, MD, PhD, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 52018
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis; YiJinJing Exercise; Hand Function; Randomized Controlled Trial
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yi Jin Jing exercise (Experimental): Yi Jin Jing exercise three times per week for 12 weeks. Each exercise lasts an hour and consists of three fundamental Yijinjing exercises.
  Interventions: Behavioral: Yi Jin Jing exercise
- Routine care (No Intervention): routine joint rehabilitation guidance, such as joint energy conservation and joint protection, basic daily activities without additional exercise.

INTERVENTIONS:
Behavioral: Yi Jin Jing exercise — Yi Jin Jing of The General Administration of Sport of China, which consists of twelve operational processes as the standard intervention
  Arms: Yi Jin Jing exercise

SUMMARY:
This study is a single-blinded, randomized, parallel controlled trial.The purpose of this experiment is to confirm how "Yijinjing" treatment affects hand function, handgrip strength, pain, morning stiffness, and mood disorder in RA patients compared to routine care.

DETAILED DESCRIPTION:
To compare the efficacy of Traditional Chinese Exercise Yijinjing and routine care on hand dysfunction,which is the clinical challenge in rheumatoid arthritis (RA), a single- centre,single-blinded, randomized controlled trial will be conducted. Sixty-six RA patients will be randomly allocated (1:1) to treatment with Yijinjing exercise or routine care. The primary outcome is a 10% improvement in the Michigan Hand Outcomes Questionnaire (MHQ) at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. meet the RA criteria by the American College of Rheumatology(ACR)/the European League Against Rheumatism(EULAR) in 2010 or the ACR in 1987
2. between the ages of 18 and 65, regardless of gender
3. DAS28≤3.2
4. joint function in grades I to II or X-ray in stages I to II
5. no use or maintenance of a stable dose of DMARDs, biological agents, or hormones within 4 weeks prior to screening
6. wrist joints or finger joints (MCP, PIP) were swollen or painful
7. tested for hand dysfunction by a professional rheumatologist
8. volunteer to participate

Exclusion Criteria:

1. Yijinjing exercise experience within the last 3 months
2. severe joint deformity (including subluxation and severe ulnar deviation) and joint ankylosis
3. other diseases affecting limb function such as trauma, fractures, infections, tumors, congenital malformations
4. present with complication diseases such as serious cardiovascular, brain, liver, lung, kidney, and hematopoietic system diseases
5. a moderate or severe cognitive impairment that unable to cooperate with the treatment
6. unwilling to join

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The Michigan Hand Outcomes Questionnaire (MHQ) | week 12
  The Michigan Hand Outcomes Questionnaire(MHQ) consists of 37 questions about six categories:(1) overall hand function; (2) activities of daily living; (3) work performance; (4) pain; (5) aesthetics; and (6) patient satisfaction with hand function, measured individually for the left and right hands. Each item is given a value between 0 and 100, with higher scores indicating superior function and higher pain ratings denoting more intense pain.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | week 12
  0 signifying "no pain" and 10 signifying "the worst intolerable agony"
The number of swollen joints, painful joints, and deformed joints | week 12
  Number of the following 28 joints: elbows, shoulders, elbow, wrists, metacarpal- phalangeal I-V, proximal interphalangeal I-V and knees which are swollen, painful or deformed.
Morning stiffness duration | week 12
  The time (minutes) of the patient's self-reported morning stiffness
Handgrip strength | week 12
  An electronic gripper will be used to assess handgrip strength (kg). Be carried out three times, the final result set by the average value.
Range of motion(ROM) | week 12
  Use a protractor to calculate the wrist flexion, dorsiflexion, ulnar deviation, radial deviation, MCP flexion, PIP flexion, and finger dorsiflexion angles(°).
Health Assessment Questionnaire Disability Index(HAQ) | week 12
  Health Assessment Questionnaire Disability Index(HAQ) contains 20 questions about daily activities such as dressing, brushing, getting up, eating, strolling, maintaining personal hygiene, touching, and holding. For each question, there is a four level that is scored from 0 (without any difficulty) to 3 (unable to do).
The Self-rating anxiety scale (SAS) | week 12
  The Self-rating Anxiety Scale (SAS) mainly consists of 20 items rated on a 4-point scale that from 0(no or little time) to 3(most or all of time).
The self-rating depression scale (SDS) | week 12
  The Self-rating Anxiety Scale (SAS) mainly consists of 20 items rated on a 4-point scale that from 0(no or little time) to 3(most or all of time).
Wrist joint ultrasonography Outcome Measures in Rheumatology (OMERACT) score | week 12
  Using the EULAR-OMERACT to classify rheumatoid arthritis synovitis and tenosynovitis.

CONTACTS AND LOCATIONS:
Overall Officials: JIANG Quan, M.D, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Chang T, Ma X, Gong X, Xia C, Jiang Q, Zhang R. Effect of traditional Chinese Yijinjing exercise on hand dysfunction in rheumatoid arthritis patients: a randomized controlled trial. Front Med (Lausanne). 2024 Nov 11;11:1454982. doi: 10.3389/fmed.2024.1454982. eCollection 2024. PMID 39588189